CLINICAL TRIAL: NCT01125358
Title: A Multicenter, Double-Blind, Placebo-Controlled Study of 3 Doses of LY2140023 in Patients With DSM-IV-TR Schizophrenia
Brief Title: A Study in Schizophrenic Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The decision to stop the trial was based on efficacy results in the overall schizophrenia participant population.
Sponsor: Denovo Biopharma LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13560; H8Y-JE-HBDC (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-05-17; First posted 2010-05-18 (Estimated); Results first posted 2021-09-14 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2012-11

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — LY 2140023

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 10 milligrams (mg) LY2140023 (Experimental)
  Interventions: Drug: LY2140023
- 80 mg LY2140023 (Experimental)
  Interventions: Drug: LY2140023
- 160 mg LY2140023 (Experimental)
  Interventions: Drug: LY2140023
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY2140023 — Administered orally, twice daily for up to 7 weeks of treatment
  Arms: 10 milligrams (mg) LY2140023; 160 mg LY2140023; 80 mg LY2140023
Drug: Placebo — Administered orally, twice daily for up to 7 weeks of treatment
  Arms: Placebo

SUMMARY:
This study is designed to compare 3 doses of LY2140023 for the treatment of schizophrenia as assessed at endpoint (up to 7 weeks) using the Clinical Utility Index (CUI), a measure of efficacy, safety, and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia as defined in the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR; APA 2000) (Disorganized, 295.10; Catatonic, 295.20; Paranoid 295.30; or Undifferentiated, 295.90) and confirmed by the Structured Clinical Interview for DSM-IV-TR (SCID)
* Non pregnant female participants who agree to use acceptable birth control
* At entry to the study must be considered moderately ill in the opinion of the investigator
* 1 year history of Schizophrenia prior to entering the study
* At study entry participants with a history of antipsychotic treatment must have a lifetime history of at least one hospitalization for the treatment of schizophrenia, not including the hospitalization required for study based on the investigator's clinical judgment. Participants who have never taken antipsychotic treatment may enter the study even without a history of hospitalization
* At study entry participants with a history of antipsychotic treatment must have a history of at least one episode of illness exacerbation requiring an intensification of treatment intervention or care in the last 2 years, not including the present episode of illness. Participants who have never taken antipsychotic treatment may enter the study without a past history of illness exacerbation and intensification of treatment in the last 2 years
* At study entry participants must have experienced an exacerbation of illness within the 4 weeks prior to entering the study, leading to an intensification of psychiatric care in the opinion of the investigator. If exacerbation occurs in participants who are presently hospitalized, the participants must not have been hospitalized longer than 60 days at entry of the study

Exclusion Criteria:

* Participated in any clinical trial with any pharmacological treatment intervention for which they received a study-related medication in the 6 months prior to visit 1
* Previously completed or withdrawn from this study, or any other study investigating LY2140023 or any predecessor molecules with glutamatergic activity
* Have any known history of receiving treatment with clozapine at any dose, as determined at baseline
* Have received treatment with a depot formulation of an antipsychotic medication within the 6 months prior entering the study
* Participants who are currently suicidal
* Females who are pregnant, nursing, or who intend to become pregnant within 30 days of completing the study
* Participants with uncorrected narrow-angle glaucoma, uncontrolled diabetes, certain diseases of the liver, renal insufficiency, untreated thyroid condition or other serious or unstable illnesses
* Have a history of one or more seizures, except for those who experienced a single simple febrile seizure between ages 6 months and 5 years
* Participants are excluded if their biological father, mother, brother, sister, or child has a history of idiopathic epilepsy
* Within 1 year of study enrollment, participants have a history of central nervous system infection, uncontrolled migraine, transient ischemic attack (TIA), or head trauma with loss of consciousness or a post-concussive
* Participants are excluded if they have a lifetime history of any of the following:

  * head trauma, stroke, or central nervous system (CNS) infection with persistent neurological deficit (focal or diffuse);
  * brain surgery;
  * an electroencephalogram with paroxysmal (epileptiform) activity, or
  * brain structural lesion, including developmental abnormalities, as determined by examination or previous neuroimaging studies that are consistent with a diagnosable neurological disease or syndrome
* Electroconvulsive therapy (ECT) within 3 months of entering the study or who will have ECT at any time during the study
* Leukopenia
* Medical history of Human Immunodeficiency Virus positive (HIV+) status
* Higher than normal blood prolactin levels
* Certain electrocardiogram results

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2010-05; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY(1-877-285-4559) or 1-317-615-4459 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (21):
- Japan (12):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aichi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kanagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kumamoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kyoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nagano
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nagasaki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saga
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toyama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yamaguchi
- South Korea (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Goyang-si
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Incheon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Naju
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Suwon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yŏngin
- Taiwan (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Changhua
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hsinchu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taipei

REFERENCES:
- [Derived] Kinon BJ, Millen BA, Zhang L, McKinzie DL. Exploratory analysis for a targeted patient population responsive to the metabotropic glutamate 2/3 receptor agonist pomaglumetad methionil in schizophrenia. Biol Psychiatry. 2015 Dec 1;78(11):754-62. doi: 10.1016/j.biopsych.2015.03.016. Epub 2015 Mar 19. PMID 25890643

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study consisted of a 1-week placebo lead-in period and a 6-week randomized, double-blind treatment period. Placebo responder is defined as ≥25% improvement in Positive and Negative Syndrome Scale (PANSS) Total Score from the start of placebo lead-in period to the end of placebo lead-in period.
Groups:
- 10 mg LY2140023: 5 milligrams (mg) of LY2140023 orally, twice daily for 6 weeks.
- 80 mg LY2140023: 40 mg of LY2140023 orally, twice daily for 6 weeks.
- 160 mg LY2140023: 80 mg of LY2140023 orally, twice daily for 6 weeks.
- Placebo: Placebo orally, twice daily for 6 weeks.
Period: Overall Study
Arm/Group | 10 mg LY2140023 | 80 mg LY2140023 | 160 mg LY2140023 | Placebo
Started | 21 | 21 | 20 | 20
Received at Least 1 Dose of Study Drug | 21 | 21 | 20 | 20
Placebo Responder | 1 | 0 | 0 | 0
Completed | 9 | 17 | 11 | 12
Not Completed | 12 | 4 | 9 | 8
Not completed — Adverse Event | 3 | 0 | 0 | 2
Not completed — Perceived Lack of Efficacy | 6 | 3 | 7 | 4
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — Sponsor Decision | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 2 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: All Randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | 10 mg LY2140023 | 80 mg LY2140023 | 160 mg LY2140023 | Placebo | Total
Number analyzed (Participants) | 21 | 21 | 20 | 20 | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.99 (10.98) | 42.03 (10.41) | 43.16 (10.33) | 38.34 (9.91) | 41.14 (10.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 9 | 10 | 40
  Male | 10 | 11 | 11 | 10 | 42
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 21 | 21 | 20 | 20 | 82
Region of Enrollment [Number; unit: participants]
  Taiwan | 1 | 2 | 1 | 1 | 5
  Japan | 18 | 16 | 17 | 17 | 68
  Korea, Republic of | 2 | 3 | 2 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: Clinical Utility Index (CUI)
Description: CUI measures the efficacy (response), tolerability (time on treatment) and safety [incidence of adverse events (AEs)] by quantifying these 3 attributes and provides a single metric for overall treatment outcome. Each component is given a score ranging from 0 to 5. The CUI Total Score is the sum of the 3 items and ranges from 0 to 15. The greater the CUI Total Score, the more effective the treatment. If a participant experiences a drug-related seizure/death, the safety component is given a score of 0 resulting in an overall CUI Total Score of 0. Analysis of variance (ANOVA) was used to calculate Least Squares (LS) mean and standard error. LS mean values were controlled for treatment, gender and pooled investigators.
Time Frame: Baseline through Week 6
Population: All participants who received at least 1 dose of study drug and had CUI Total Score measurement at Week 6.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 10 mg LY2140023 | 80 mg LY2140023 | 160 mg LY2140023
Number analyzed (Participants) | 21 | 21 | 20
units on a scale | 8.30 (0.54) | 10.32 (0.52) | 9.27 (0.55)
Statistical Analysis 1: Comparison: 10 mg LY2140023 vs 80 mg LY2140023; Test type: Superiority or Other; Multiple Comparisons with The Best (MCB); LS mean difference = LS mean of 10 mg LY2140023 - LS mean of 80 mg LY2140023; LS Mean Differences = -2.02, 90% CI 2-sided [-3.37 to 0.00]
Statistical Analysis 2: Comparison: 80 mg LY2140023 vs 160 mg LY2140023; Test type: Superiority or Other; Multiple Comparison with The Best (MCB); LS mean difference = LS mean of 160 mg LY2140023 - LS mean of 80 mg LY2140023; LS Mean Differences = -1.05, 90% CI 2-sided [-2.42 to 0.32]

2. Secondary Outcome: Change From Baseline to Week 6 Endpoint in the Positive and Negative Syndrome Scale (PANSS) Total Score, Positive Score, Negative Score, and Psychopathology Subscale
Description: The PANSS consists of 30 items and 3 subscales designed to measure severity of psychopathology in schizophrenia. The PANSS Positive Subscale and the PANSS Negative Subscale each contain 7 items, and the remaining 16 items make up the PANSS General Psychopathology Subscale. Each item is rated from 1 (symptom not present) to 7 (symptom extremely severe). The PANSS Total Score is the sum of the 30 items (range from 30 to 210). The PANSS Positive Subscale and PANSS Negative Subscale scores each range from 7 to 49. The PANSS General Psychopathology Subscale score ranges from 16 to 112. Higher scores indicate greater severity of illness. The Mixed Model Repeated Measures (MMRM) analysis was used to calculate Least Squares (LS) mean and 95% confidence interval. LS mean values were controlled for baseline, treatment, gender, pooled investigator, visit, treatment*visit and baseline*visit.
Time Frame: Baseline, Week 6
Population: All randomized participants who received at least 1 dose of study drug, had a baseline and at least 1 post-baseline PANSS measurement. Placebo responder (defined as ≥25% improvement in the PANSS Total Score from the start of placebo lead-in period to the end of placebo lead-in period) was excluded from the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | 10 mg LY2140023 | 80 mg LY2140023 | 160 mg LY2140023 | Placebo
Number analyzed (Participants) | 19 | 21 | 20 | 20
units on a scale
  PANSS Total Score | -0.49 [-12.37 to 11.40] | -2.56 [-12.32 to 7.20] | 1.40 [-9.64 to 12.44] | 9.35 [-1.80 to 20.51]
  PANSS Positive Subscore (n=19, 21, 20, 20) | 0.33 [-2.80 to 3.45] | -2.30 [-4.90 to 0.30] | -0.05 [-2.93 to 2.82] | 1.93 [-1.00 to 4.85]
  PANSS Negative Subscore | 0.23 [-3.20 to 3.67] | -0.22 [-3.03 to 2.58] | 0.33 [-2.84 to 3.50] | 2.70 [-0.50 to 5.90]
  PANSS General Psychopathology Subscore | -0.88 [-7.05 to 5.30] | -0.31 [-5.35 to 4.72] | 1.18 [-4.59 to 6.94] | 4.79 [-1.03 to 10.60]
Statistical Analysis 1: Comparison: 10 mg LY2140023 vs Placebo; Test type: Superiority or Other; p = 0.222, MMRM — P-value is for PANSS Total Score; LS Mean Differences = -9.84, 95% CI 2-sided [-25.80 to 6.12], Standard Error of Mean 7.96
Statistical Analysis 2: Comparison: 80 mg LY2140023 vs Placebo; Test type: Superiority or Other; p = 0.105, MMRM — P-value is for PANSS Total Score; LS Mean Differences = -11.91, 95% CI 2-sided [-26.42 to 2.60], Standard Error of Mean 7.22
Statistical Analysis 3: Comparison: 160 mg LY2140023 vs Placebo; Test type: Superiority or Other; p = 0.308, MMRM — P-value is for PANSS Total Score; LS Mean Differences = -7.96, 95% CI 2-sided [-23.46 to 7.55], Standard Error of Mean 7.73
Statistical Analysis 4: Comparison: 10 mg LY2140023 vs Placebo; Test type: Superiority or Other; p = 0.441, MMRM — P-value is for PANSS Positive Subscore; LS Mean Differences = -1.60, 95% CI 2-sided [-5.74 to 2.54], Standard Error of Mean 2.06
Statistical Analysis 5: Comparison: 80 mg LY2140023 vs Placebo; Test type: Superiority or Other; p = 0.030, MMRM — P-value is for PANSS Positive Subscore; LS Mean Differences = -4.22, 95% CI [-8.01 to -0.44], Standard Error of Mean 1.88
Statistical Analysis 6: Comparison: 160 mg LY2140023 vs Placebo; Test type: Superiority or Other; p = 0.323, MMRM — P-value is for PANSS Positive Subscore; LS Mean Differences = -1.98, 95% CI 2-sided [-5.96 to 2.01], Standard Error of Mean 1.98
Statistical Analysis 7: Comparison: 10 mg LY2140023 vs Placebo; Test type: Superiority or Other; p = 0.285, MMRM — P-value is for PANSS Negative Subscore; LS Mean Differences = -2.46, 95% CI 2-sided [-7.05 to 2.12], Standard Error of Mean 2.28
Statistical Analysis 8: Comparison: 80 mg LY2140023 vs Placebo; Test type: Superiority or Other; p = 0.166, MMRM — P-value is for PANSS Negative Subscore; LS Mean Differences = -2.92, 95% CI 2-sided [-7.10 to 1.26], Standard Error of Mean 2.07
Statistical Analysis 9: Comparison: 160 mg LY2140023 vs Placebo; Test type: Superiority or Other; p = 0.286, MMRM — P-value is for PANSS Negative Subscore; LS Mean Differences = -2.37, 95% CI 2-sided [-6.79 to 2.05], Standard Error of Mean 2.20
Statistical Analysis 10: Comparison: 10 mg LY2140023 vs Placebo; Test type: Superiority or Other; p = 0.177, MMRM — P-value is for PANSS General Psychopathology Subscore; LS Mean Differences = -5.67, 95% CI 2-sided [-13.96 to 2.63], Standard Error of Mean 4.14
Statistical Analysis 11: Comparison: 80 mg LY2140023 vs Placebo; Test type: Superiority or Other; p = 0.178, MMRM — P-value is for PANSS General Psychopathology Subscore; LS Mean Differences = -5.10, 95% CI 2-sided [-12.60 to 2.40], Standard Error of Mean 3.74
Statistical Analysis 12: Comparison: 160 mg LY2140023 vs Placebo; Test type: Superiority or Other; p = 0.377, MMRM — P-value is for PANSS General Psychopathology Subscore; LS Mean Differences = -3.61, 95% CI 2-sided [-11.72 to 4.51], Standard Error of Mean 4.05

3. Secondary Outcome: Change From Baseline to Week 6 Endpoint in the Clinical Global Impression-Severity Scale (CGI-S)
Description: The CGI-S instrument is used to record the severity of mental illness at the time of assessment. The score ranges from 1 (normal, not at all ill) to 7 (among the most extremely ill). Higher scores indicate greater severity of illness. The Mixed Model Repeated Measures (MMRM) analysis was used to calculate Least Squares (LS) mean and 95% confidence interval. LS mean values were controlled for baseline, treatment, gender, pooled investigator, visit, treatment*visit and baseline*visit.
Time Frame: Baseline, Week 6
Population: All randomized participants who received at least 1 dose of study drug, had a baseline and at least 1 post-baseline CGI-S measurement. Placebo responder (defined as ≥25% improvement in the PANSS Total Score from the start of placebo lead-in period to the end of placebo lead-in period) was excluded from the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | 10 mg LY2140023 | 80 mg LY2140023 | 160 mg LY2140023 | Placebo
Number analyzed (Participants) | 19 | 21 | 20 | 20
units on a scale | 0.62 [-0.11 to 1.34] | -0.49 [-1.09 to 0.11] | 0.14 [-0.52 to 0.81] | -0.25 [-0.93 to 0.42]
Statistical Analysis 1: Comparison: 10 mg LY2140023 vs Placebo; Test type: Superiority or Other; p = 0.077, MMRM; LS Mean Differences = 0.87, 95% CI 2-sided [-0.10 to 1.83], Standard Error of Mean 0.48
Statistical Analysis 2: Comparison: 80 mg LY2140023 vs Placebo; Test type: Superiority or Other; p = 0.592, MMRM; LS Mean Differences = -0.24, 95% CI 2-sided [-1.12 to 0.65], Standard Error of Mean 0.44
Statistical Analysis 3: Comparison: 160 mg LY2140023 vs Placebo; Test type: Superiority or Other; p = 0.395, MMRM; LS Mean Differences = 0.39, 95% CI 2-sided [-0.53 to 1.32], Standard Error of Mean 0.46

4. Secondary Outcome: Change From Baseline to Week 6 Endpoint in the 16-item Negative Symptoms Assessment (NSA-16)
Description: The NSA-16 scale is used to help clinicians rate behaviors (not psychopathology) commonly associated with negative symptoms of schizophrenia. The scale rates participants on 16 "anchors". Each item ("anchor") is rated from 1 (better) to 6 (worse). The NSA-16 Total Score is the sum of the 16 specific items and ranges from 16 to 96. Higher scores indicate greater severity of illness. The Mixed Model Repeated Measures (MMRM) analysis was used to calculate Least Squares (LS) mean and 95% confidence interval. LS mean values were controlled for baseline, treatment, gender, pooled investigator, visit, treatment*visit and baseline*visit.
Time Frame: Baseline, Week 6
Population: All randomized participants who received at least 1 dose of study drug, had a baseline and at least 1 post-baseline NSA-16 Total Score measurement. Placebo responder (defined as ≥25% improvement in the PANSS Total Score from the start of placebo lead-in period to the end of placebo lead-in period) was excluded from the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | 10 mg LY2140023 | 80 mg LY2140023 | 160 mg LY2140023 | Placebo
Number analyzed (Participants) | 13 | 17 | 14 | 13
units on a scale | 3.42 [-3.38 to 10.22] | -0.40 [-6.41 to 5.60] | -6.31 [-13.16 to 0.53] | -1.22 [-7.76 to 5.33]
Statistical Analysis 1: Comparison: 10 mg LY2140023 vs Placebo; Test type: Superiority or Other; p = 0.306, MMRM; LS Mean Differences = 4.64, 95% CI 2-sided [-4.37 to 13.65], Standard Error of Mean 4.49
Statistical Analysis 2: Comparison: 80 mg LY2140023 vs Placebo; Test type: Superiority or Other; p = 0.849, MMRM; LS Mean Differences = 0.82, 95% CI 2-sided [-7.74 to 9.38], Standard Error of Mean 4.26
Statistical Analysis 3: Comparison: 160 mg LY2140023 vs Placebo; Test type: Superiority or Other; p = 0.259, MMRM; LS Mean Differences = -5.09, 95% CI [-14.05 to 3.86], Standard Error of Mean 4.46

5. Secondary Outcome: The Number of Participants With Treatment-Emergent Suicidal Ideation and Behavior Based on the Columbia Suicide Severity Rating Scale (C-SSRS)
Description: Columbia Suicide Rating Scale (C-SSRS) captures occurrence, severity, and frequency of suicide-related thoughts and behaviors. Suicidal ideation: a "yes" answer to any one of 5 suicidal ideation questions: wish to be dead, and 4 different categories of active suicidal ideation. Suicidal behavior: a "yes" answer to any of 5 suicidal behavior questions: preparatory acts or behavior, aborted attempt, interrupted attempt, non-fatal suicide attempt, and completed suicide. The number of participants with statistically significant changes of the C-SSRS was the number of participants with a treatment-emergent suicidal ideation and behavior (an increase in suicidal behavior or ideation over lead-in baseline.)
Time Frame: Baseline up to Week 6
Population: All randomized participants who received at least 1 dose of study drug and had a baseline and at least 1 post-baseline C-SSRS measurements.
Measure: Number; unit: participants
Arm/Group | 10 mg LY2140023 | 80 mg LY2140023 | 160 mg LY2140023 | Placebo
Number analyzed (Participants) | 20 | 21 | 20 | 20
participants
  Treatment-Emergent Suicidal Ideation | 1 | 1 | 2 | 1
  Treatment-Emergent Suicidal Behavior | 0 | 0 | 0 | 0

6. Secondary Outcome: Percentage of Participants Who Discontinued (Rate of Discontinuation)
Description: Rate of discontinuation was calculated as the number of participants who discontinued from study due to any reason divided by the total number of participants who received study drug, then multiplied by 100.
Time Frame: Baseline through Week 6
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | 10 mg LY2140023 | 80 mg LY2140023 | 160 mg LY2140023 | Placebo
Number analyzed (Participants) | 21 | 21 | 20 | 20
percentage of participants | 57.1 | 19.0 | 45.0 | 40.0
Statistical Analysis 1: Comparison: 10 mg LY2140023 vs Placebo; Test type: Superiority or Other; p = 0.354, Fisher Exact
Statistical Analysis 2: Comparison: 80 mg LY2140023 vs Placebo; Test type: Superiority or Other; p = 0.181, Fisher Exact
Statistical Analysis 3: Comparison: 160 mg LY2140023 vs Placebo; Test type: Superiority or Other; p > 0.999, Fisher Exact

ADVERSE EVENTS:
Arm/Group | 10 mg LY2140023 | 80 mg LY2140023 | 160 mg LY2140023 | Placebo
Serious Adverse Events (participants affected / at risk) | 1/21 | 2/21 | 0/20 | 2/20
Other Adverse Events (participants affected / at risk) | 13/21 | 13/21 | 12/20 | 9/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 10 mg LY2140023 (N=21) | 80 mg LY2140023 (N=21) | 160 mg LY2140023 (N=20) | Placebo (N=20)
Psychomotor hyperactivity (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Schizophrenia (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 10 mg LY2140023 (N=21) | 80 mg LY2140023 (N=21) | 160 mg LY2140023 (N=20) | Placebo (N=20)
Visual impairment (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 2 (3) | 1 (1)
Oral disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retching (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 4 (4) | 1 (1) | 2 (2)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinea pedis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin unconjugated increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood prolactin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood uric acid increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Affect lability (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Affective disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Delusion (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Schizophrenia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0/11 (0) | 1/10 (1) | 0/9 (0) | 0/10 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hair colour changes (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days